CLINICAL TRIAL: NCT03475862
Title: A Randomized, Double-Blind, Placebo-Controlled, Double-Dummy, Single-Dose,4-Way Crossover Study With Exploratory Fifth Treatment to Determine the Relative Nasal Abuse Potential of PTI-821 (Oxycodone Extended-Release Capsules)
Brief Title: Nasal Human Abuse Potential of PTI-821
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pain Therapeutics (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Organization: PainT (Unknown)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: PTI-821-C08
Record Dates: First submitted 2018-03-07; First posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Opioid Abuse Nondependent
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Intervention Model Description: 4-way single-dose crossover with an exploratory 5th treatment arm
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, double-dummy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- PTI-821 Manipulated (Experimental): oxycodone 40 mg capsule
  Interventions: Drug: PTI-821 capsule Manipulated
- Oxycodone (Active Comparator): Oxycodone 40 mg IR tablet crushed
  Interventions: Drug: Oxycodone
- OxyContin (Active Comparator): Oxycodone ER 40 mg tablet crushed
  Interventions: Drug: OxyContin
- Placebo (Placebo Comparator): Matching placebos for experimental and active comparator arms
  Interventions: Other: Placebo
- PTI-821 Non-manipulated (Experimental): Oxycodone 40 mg non-manipulated
  Interventions: Drug: PTI-821 Non-manipulated

INTERVENTIONS:
Drug: PTI-821 capsule Manipulated — PTI-821 (oxycodone) 40 mg extended release capsule
  Arms: PTI-821 Manipulated
Drug: PTI-821 Non-manipulated — PTI-821 (oxycodone) 40 mg capsule extended release capsule
  Arms: PTI-821 Non-manipulated
Drug: OxyContin — Crushed OxyContin (oxycodone) extended-release 40 mg tablet
  Arms: OxyContin
Other: Placebo — Matching placebos for PTI-821 and oxycodone IR
  Arms: Placebo
Drug: Oxycodone — Crushed oxycodone 40 mg immediate release tablet
  Arms: Oxycodone

SUMMARY:
The study will evaluate the human abuse liability of PTI-821 (oxycodone extended-release capsules) when administered nasally compared to crushed oxycodone IR tablets and crushed OxyContin tablets, also administered nasally.

DETAILED DESCRIPTION:
The nasal human abuse liability of PTI-821 will be compared to oxycodone IR using pharmacokinetic and pharmacodynamic assessments. A comparison to OxyContin will be dose using pharmacokinetic assessments.

ELIGIBILITY:
Inclusion Criteria::

* Healthy male and/or female subjects between the ages of 18 and 55 years,
* Subject is a recreational opioid user who is NOT dependent on opioids
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and body weight > 50 kg (110lbs).
* Evidence of a personally signed and dated informed consent document
* Subjects must be willing and able to comply with study procedures.
* Females who are physically incapable of childbearing, or practicing an acceptable method of birth control. Acceptable methods of birth control include surgical sterilization, hormonal contraceptives, or double-barrier methods (condom or diaphragm with a spermicidal agent or intrauterine device).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Diagnosis of substance and/or alcohol dependence (excluding caffeine and nicotine).
* Has participated in, is currently participating in, or is seeking treatment for substance- and/or alcohol-related disorders (excluding nicotine and caffeine).
* Has a positive urine drug screen (UDS) excluding tetrahydrocannabinol (THC) at Screening and the admission for Qualification Phase.
* Has a positive alcohol breath test at Screening or upon admission to the study center for the Qualification Phase.
* Has any history of a condition in which an opioid is contraindicated
* History of sleep apnea in the past 5 years that has not been resolved.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject unsuitable for entry into this study.
* Positive test for Hepatitis B, Hepatitis C, or HIV at Screening.
* Allergy or history of hypersensitivity to naloxone hydrochloride (HCl), oxycodone HCl, other opioids, and/or lactose.
* Any condition possibly affecting drug absorption.
* Physical (eg, constricted or collapsed veins) or mental obstruction (ie, phobia) that would prevent serial blood sample collection.
* Clinically significant illness in the judgment of the investigator within 30 days before Screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first treatment during the Qualification Period (Visit 2), if longer than 30 days.
* Screening BP > 140 mm Hg (systolic) or > 90 mm Hg (diastolic) following at least 5 minutes of rest. If BP is > 140 mm Hg (systolic) or > 90 mm Hg (diastolic), the BP should be repeated two more times and the average of the three BP values should be used to determine the subject's eligibility.
* Pregnant females; breastfeeding females; males and females of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for 28 days after the last dose of study medication. Urine pregnancy tests must be collected and confirmed negative prior to dosing upon admission.
* Is currently taking a drug for a medical condition or a nutraceutical that poses a safety risk when administered with an opioid, cannot be safely withdrawn at Screening for the duration of the study, and/or will adversely affect the PD and safety assessments required by the study. Examples include antihypertensive agents, drugs for seizures, and diabetes medications. Hormonal contraceptives (oral, injected, intrauterine, transdermal or implanted) are allowed in this study provided the subject remains on the same treatment throughout the entire study and has been using that hormonal contraceptive for an adequate period of time to ensure effectiveness. Limited use of non-prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the investigator. As an exception, acetaminophen may be used at doses of 1 g/day.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 30 days prior to dosing.
* Unwilling or unable to comply with the procedures described in this protocol.
* Unwilling to be searched (including personal effects) for illicit substances before admission to the study center.
* Subject is a heavy smoker (> 20 cigarettes per day on average in the past 30 days prior to Screening), chews tobacco, uses nicotine-containing products (including nicotine transdermal patches), and/or is unable to abstain from smoking for at least 10 hours during any day.
* Current pending legal charges or currently on probation.
* Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are PTI employees directly involved in the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Drug Liking Emax | Intervals from 0.5 hours to 12 hours post dose
  Peak effect for drug liking based on bipolar visual analog scale from 0-100 where 0 is most negative response, 50 is neutral, and 100 is most positive response.

SECONDARY OUTCOMES:
Take Drug Again | 12 and 25 hours
  Desire to take drug again if offered based on bipolar visual analog scale from 0-100 where o is most negative response, 50 is neutral, and 100 is the most positive response.
Drug effects questionnaire | Intervals from 0.5 hours to 12 hours post dose
  Assesses various drug effects such as good drug effects, bad drug effects, high and nausea/dizziness
Peak Plasma Concentration (Cmax) | Intervals from 15 minutes to 24 hours post-dose
  Maximum plasma concentration
Area under the plasma concentration versus time curve | Intervals from 15 minutes to 24 hours post-dose
  Amount of drug absorbed at various timepoints
Time to maximum plasma concentration (Tmax) | Intervals from 15 minutes to 24 hours post-dose
  The time intervals from the first dose to the peak plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Webster, MD, Principal Investigator — PRA Health Sciences
Locations (1):
- PRA-EDS, Salt Lake City, Utah, United States